CLINICAL TRIAL: NCT03363555
Title: An Open-Label, Single Arm, Multi-Center, Phase 2 Study of PD-1 Antibody SHR-1210 in Subjects With Relapsed or Refractory Extranodal NK/T Cell Lymphoma
Brief Title: SHR-1210 in Patients With Relapsed or Refractory Extranodal NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-205
Record Dates: First submitted 2017-11-29; First posted 2017-12-06 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 (Experimental): SHR-1210 injection, 200 mg/dose, intravenous infusion within 20-60 minutes.
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — A humanized monoclonal immunoglobulin.

SUMMARY:
This is an open-label, multi-center, nonrandomized, Phase 2 study to evaluate efficacy and safety of SHR-1210 in subjects with relapsed or refractory extranodal NK/T cell lymphoma.Efficacy will be assessed every 8 weeks according to 2014 Lugano criteria.Safety evaluations (both clinical and laboratory) are performed at baseline, before each study treatment, and throughout the study.

DETAILED DESCRIPTION:
The primary objective of this phase 2 study is to assess objective response rate of SHR-1210 in patients with relapsed or refractory extranodal NK/T cell lymphoma. The secondary objective is to observe time to response,progression free survival rate at 2 years,overall survival rate at 2 years，safety and immunogenicity of SHR-1210 in relapsed or refractory extranodal NK/T cell lymphoma.The relationship of PD-L1 expression in tumor tissue and EBV-DNA copies in blood to SHR-1210 efficacy in these patients would also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed extranodal NK/T cell lymphoma;
2. Relapsed or refrsctory cHL and received L-asparaginase based chemotherapy.
3. Subjects enrolled have measurable lesion(s) according to Lugano 2014 criteria
4. Need to provide ≥5 tumor tissue sections for detection.
5. ECOG performance status of 0 or 1;
6. Life expectancy ≥ 12 weeks.;
7. Adequate laboratory parameters during the screening period as evidenced by the following:

   1. Absolute neutrophil count ≥ 1.0× 109/L ;
   2. Platelets ≥ 75 × 109/L;
   3. Hemoglobin ≥ 8.0 g/dL;
   4. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), ALT and AST ≤ 2.5×ULN
   5. Serum Creatinine ≤1.25×ULN or Creatinine clearance≥45 mL/min;
   6. Coagulation function index：INR ≤1.5×ULN，APTT≤1.5×ULN
8. Women of childbearing potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 60 days after receiving the last dose of study treatment. Women of childbearing potential with pregnancy test negative within 7days before entering the group and not in in lactation; Male subjects with WOCBP partner should receive Surgical sterilization orconsent to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 120 days after receiving the last dose of study treatment.
9. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. invasive NK cell leukemia or precursor NK cell tumor
2. Known central nervous system lymphoma
3. Haemophilus cell syndrome at diagnosis
4. Large lung vessels were involved
5. History and complication

   1. Recieved anti-tumor vaccines or other anti-tumor therapy with immune stimulation within 3 months.
   2. Prior exposure to any PD-1/PD-L1/PD -L 2 or CTLA -4 antibody .
   3. Participating in other clinical studies or less than 4 weeks before the end of a clinical trial;
   4. Active, known or suspected autoimmune disease. Subjects who were in a stable state without systemic immunosuppressive therapy were admitted.
   5. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic corticosteroids > 10mg.
   6. Known and suspicion of interstitial pneumonia
   7. Other active malignancies that required treating.
   8. Received chemotherapy, radiotherapy,immunotherapy, including topical therapy within 4 weeks. Previous anti-tumor therapy related adverse reactions (except trichomadesis) did not recover to CTCAE ≤1.
   9. Prior allo-HSCT.
   10. ASCT within 90 days.
   11. Impact of major surgery or severe trauma had been eliminated for less than 14 days.
   12. Active pulmonary tuberculosis.
   13. Severe acute or chronic infection requiring systemic therapy.
   14. Suffering from heart failure (New York Heart Association standard III or IV) and given appropriate medical treatment.Uncontrolled coronary artery disease and arrhythmia. History of myocardial infarction within 6 months.
6. laboratory test

   1. known HIV positive or known AIDS.
   2. Untreated active hepatitis; Hepatitis B and hepatitis C infection in common.
7. Other factors that may lead to the study termination, such as severe disease or abnormal laboratory tests or family or social factors affecting subjects safety or test data and sample collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
objective response rate | from first patient first visit to 6 month after last patient first visit
  rate of subjects achieved complete response plus partial response in all evaluable subjects

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No